CLINICAL TRIAL: NCT03219047
Title: A Pilot Study Evaluating Xenografts to Personalize Therapies (PDX) in Relapsed Mantle Cell Lymphoma to Optimize Response: The EXPLORE Trial
Brief Title: Patient-Derived Xenografts in Personalizing Treatment for Patients With Relapsed/Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0051; NCI-2018-01117 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0051 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Practice Guidelines as Topic; Standard of Care; ibrutinib; Precision Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 2 (Co-trial cohort) (Experimental): Patients receive ibrutinib at standard dose and schedule through an ongoing MD Anderson clinical trial. Patients that respond to ibrutinib but experience relapse or disease progression receive treatment based on the results of the PDX models as in Cohort 1 if they are available. Patients who experience relapse after treatment with ibrutinib are moved to Cohort I if the PDX models are not ready.
  Interventions: Other: Best Practice; Drug: Ibrutinib; Other: Patient Derived Xenograft; Other: Personalized Medicine
- Cohort I (Traditional cohort) (Experimental): Patients who have previously received ibrutinib, acalabrutinib, PI3K inhibitor ACP-319, or BTK inhibitor BGB-3111 receive treatment through ongoing clinical trials at MD Anderson or standard of care. At the same time, previously collected tissue is used to develop PDX models and suitable drugs/regimens are tested in the PDX models. Patients then receive treatment based on the results of the PDX models through another clinical trial or standard of care.
  Interventions: Other: Best Practice; Other: Patient Derived Xenograft; Other: Personalized Medicine

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Drug: Ibrutinib — Given at standard dose and schedule
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
  Arms: Cohort 2 (Co-trial cohort)
Other: Patient Derived Xenograft — Xenograft developed
  Other Names: Patient-Derived Xenograft; Patient-Derived Xenograft Model; PDTX; PDX
Other: Personalized Medicine — Receive treatment based on the results of the PDX models

SUMMARY:
This early phase I pilot trial studies how well patient-derived xenografts work in personalizing treatment for patients with mantle cell lymphoma that has come back (relapsed) or that isn't responding to treatment (refractory). Xenograft models involve taking a piece of tissue from a tumor that was previously collected and putting that tissue inside of a mouse in the laboratory. This allows the tumor to grow in the mouse so that researchers can test the effects of certain drugs. If the drugs have an effect on the tumor(s) in the mice, patients may receive that treatment for mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility in the patients treated with the patient-derived xenografts (PDX)-directed therapies in both cohorts (cohort 1 and cohort 2).

II. To establish mouse xenografts from the mantle cell lymphoma (MCL) tissue samples of patients with relapsed MCL.

III. To determine the activity of a panel of anticancer drugs consistent with the patient's clinical history against these MCL cells in vitro.

IV. To test the best selected in vitro options in the PDX model to create a profile, in rank order based on the efficacy of best 3-5 options, of individualized patient treatment options.

V. To determine the feasibility of predicting the patient's response to therapy using a PDX-based strategy.

VI. To define susceptibility and resistance determinants to the drugs in xenografted tumors.

SECONDARY OBJECTIVES:

I. To determine the objective response (OR) rate (complete + partial responses).

II. To determine safety and toxicity. III. To determine progression-free survival (PFS).

EXPLORATORY OBJECTIVES:

I. To correlate detected gene mutations and changes in ribonucleic acid (RNA) and/or protein expression with treatment responses.

OUTLINE: patients are assigned to 1 of 2 cohorts.

COHORT 1 (TRADITIONAL COHORT): Patients who have previously received ibrutinib, acalabrutinib, PI3K inhibitor ACP-319, or BTK inhibitor BGB-3111 receive treatment through ongoing clinical trials at MD Anderson or standard of care. At the same time, previously collected tissue is used to develop PDX models and suitable drugs/regimens are tested in the PDX models. Patients then receive treatment based on the results of the PDX models through another clinical trial or standard of care.

COHORT 2 (CO-TRIAL COHORT): Patients receive ibrutinib at standard dose and schedule through an ongoing MD Anderson clinical trial. Patients that respond to ibrutinib but experience relapse or disease progression receive treatment based on the results of the PDX models as in Cohort 1 if they are available. Patients who experience relapse after treatment with ibrutinib are moved to Cohort I if the PDX models are not ready.

ELIGIBILITY:
Inclusion Criteria:

* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Confirmed MCL tissue diagnosis.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Patients must have relapsed/progressed after any therapy for MCL.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Patients must be willing to allow residual tissue to be collected for both in vitro, in vivo (PDX) testing and molecular profiling.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Patients must have bi-dimensional measurable disease as per Lugano criteria (bone marrow or gastrointestinal [GI] only involvement is acceptable).
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Disease free of other prior malignancies of >= 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy) or not actively being treated, with a life expectancy > 2 years.
* FOR TISSUE COLLECTION TO ESTABLISH PDX (PART 1): Reasonable expectation that the patient can wait 3-6 months for generation of PDX data for subsequent treatment selection.
* FOR PDX-GUIDED THERAPY THROUGH ONGOING TRIALS AT MD ANDERSON OR OFF-PROTOCOL WITH STANDARD OF CARE (PART 2): The patient PDXs must have generated informative mouse xenograft data during Part 1 to participate in Part 2.
* FOR PDX-GUIDED THERAPY THROUGH ONGOING TRIALS AT MD ANDERSON OR OFF-PROTOCOL WITH STANDARD OF CARE (PART 2): The patient condition remains suitable for the selected therapy. If the patient receives prior therapy with a given agent (X) and progressed, but the testing in Part 1 found this agent to be effective in a combination, the patient remains eligible for this combination that includes agent X.
* FOR PDX-GUIDED THERAPY THROUGH ONGOING TRIALS AT MD ANDERSON OR OFF-PROTOCOL WITH STANDARD OF CARE (PART 2): Patients should ideally have bi-dimensional measurable disease (leukemia phase only, bone marrow only, splenomegaly only, or GI involvement only is acceptable).
* FOR PDX-GUIDED THERAPY THROUGH ONGOING TRIALS AT MD ANDERSON OR OFF-PROTOCOL WITH STANDARD OF CARE (PART 2): Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. Men must agree not to father a child and agree to use a condom if his partner is of child-bearing potential.
* FOR PDX-GUIDED THERAPY THROUGH ONGOING TRIALS AT MD ANDERSON OR OFF-PROTOCOL WITH STANDARD OF CARE (PART 2): Patients must have adequate organ function for drugs(s) or combination being utilized (dependent on the drug[s] being given).

Exclusion Criteria:

* Any serious medical condition that places the patient at unacceptable risk and/or would prevent the subject from signing the informed consent form. Examples include but are not limited to uncontrolled hypertension, uncontrolled diabetes mellitus, active /symptomatic coronary artery disease, active infection, active hemorrhage, and psychiatric illness.
* Pregnant or breastfeeding females.
* Known human immunodeficiency virus (HIV) infection. Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation.
* The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL with a life expectancy < 2 years.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months at the time of consent or any class 3 (moderate) or 4 (severe) cardiac disease defined by the New York Heart Association classification.
* Prior chemotherapy within 3 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, major surgery within 4 weeks or vaccination with live attenuated vaccines within 4 weeks of the first dose of study drug.
* THE PATIENT IS INELIGIBLE TO PARTICIPATE IN PART 2 IF ANY OF THE FOLLOWING OCCUR: PDX data are non-informative.
* THE PATIENT IS INELIGIBLE TO PARTICIPATE IN PART 2 IF ANY OF THE FOLLOWING OCCUR: Tumors do not engraft in the mice or do not respond to any of the selected agents.
* THE PATIENT IS INELIGIBLE TO PARTICIPATE IN PART 2 IF ANY OF THE FOLLOWING OCCUR: In Cohort 2, if disease progression occurs before Part 1 data are available, then they will be transferred to Cohort 1.
* THE PATIENT IS INELIGIBLE TO PARTICIPATE IN PART 2 IF ANY OF THE FOLLOWING OCCUR: Part 1 data contradict clinical judgment. The investigator should discuss with the principal investigator (PI) and use the best discretion.
* THE PATIENT IS INELIGIBLE TO PARTICIPATE IN PART 2 IF ANY OF THE FOLLOWING OCCUR: Any other exclusion criteria set forth by individual treatment protocol of the active clinical trial(s) through which patients are going to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Feasibility defined as available patient-derived xenograft (PDX) results before relapse | Up to 1 year
  This will be established if both PDX model is built successfully based on the primary tumor samples, and the results of the PDX results are available before disease relapse. We consider the study feasible if the posterior probability of feasibility rate above 30% is larger than 80% at the end of the study. The feasibility rate in each cohort will be summarized by frequency and 95% posterior credible interval.

SECONDARY OUTCOMES:
Objective response (OR) rate (complete + partial responses) | Up to 1 year
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate. Will be estimated by a Bayesian posterior credible interval, and summarized by frequency and 95% posterior credible interval.
Incidence of adverse events | Up to 1 year
  Toxicity data by type and severity will be summarized by frequency tables. Will be estimated by a Bayesian posterior credible interval, and summarized by frequency and 95% posterior credible interval.
Progression-free survival (PFS) | Up to 1 year
  The distribution of PFS will be estimated using the method of Kaplan and Meier. Cox proportional hazard regression will be employed for multivariate analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org